CLINICAL TRIAL: NCT07319338
Title: Implementing Objective Vascular Biomarkers as a Non-stigmatizing Triage Workflow for Depression in Gastroenterology Settings: a Multicenter Study Protocol for a Hybrid Effectiveness-implementation Study
Brief Title: Objective Vascular Biomarkers as Triage for Depression in Chronic Atrophic Gastritis
Status: Not yet recruiting | Type: Observational
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing Anzhen Hospital (Other); Hengshui Hospital of Traditional Chinese Medicine (Unknown); Liyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Meng Wang, Principal Investigator, China Academy of Chinese Medical Sciences
Other Study IDs: 2025-EC-KY-004; Other Identifier (Other: 2025-KY-18)
Record Dates: First submitted 2025-12-11; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Atrophic Gastritis; Depressive Symptoms; Depression; Gastrointestinal Diseases
Keywords: Vascular biomarkers; Dorsalis pedis artery ultrasound; Triage workflow; Implementation science; Stigma; Screening; Gut-brain axis
MeSH Terms: conditions — Gastritis, Atrophic; Depression; Gastrointestinal Diseases; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Chronic Atrophic Gastritis (CAG): Adults (aged 20-60 years) with histologically confirmed chronic atrophic gastritis diagnosed via upper gastrointestinal endoscopy within the past 6 months.
  Interventions: Diagnostic Test: Vascular-Psychological Triage Workflow

INTERVENTIONS:
Diagnostic Test: Vascular-Psychological Triage Workflow — Participants undergo a multimodal assessment including high-frequency ultrasound of the dorsalis pedis artery, measurement of brachial-ankle pulse wave velocity (baPWV), and completion of the PHQ-9 depression screening scale.

SUMMARY:
Depressive symptoms are highly prevalent in patients with chronic atrophic gastritis (CAG) but are frequently under-detected due to stigma and reliance on subjective questionnaires. This multicenter, cross-sectional observational study aims to validate a novel clinical triage workflow. It repurposes routine vascular assessments (specifically dorsalis pedis artery ultrasound and arterial stiffness metrics) as objective "biological entry points" to facilitate mental health referrals. The study will enroll approximately 450-520 adults with histologically confirmed CAG across four clinical centers in China. The primary objective is to determine the diagnostic accuracy of these vascular biomarkers for identifying patients with moderate-to-severe depressive symptoms (PHQ-9 score >= 10). Secondary objectives include evaluating the implementation feasibility (e.g., referral uptake, screening completion rate) of this integrated care model in routine gastroenterology practice.

DETAILED DESCRIPTION:
Current screening for depression in gastroenterology relies heavily on self-report scales, which are often limited by somatization and cultural stigma in Asian populations. This study proposes a "vascular-gut-brain" framework to bridge this service gap.

Participants will undergo a standardized multimodal assessment comprising:

* Gastrointestinal evaluation: Endoscopy and histopathology (OLGA/OLGIM staging), and symptom scoring (GSRS).

  * Peripheral vascular assessment: High-frequency ultrasound of the dorsalis pedis artery (measuring Resistive Index [RI], Pulsatility Index [PI], and waveform classification).

    * Arterial stiffness and autonomic function: Brachial-ankle pulse wave velocity (baPWV), Ankle-Brachial Index (ABI), and Heart Rate Variability (HRV).

      * Psychological assessment: PHQ-9, GAD-7, and PSQI scales.

The study employs a hybrid effectiveness-implementation design. In addition to validating the diagnostic accuracy of vascular markers, the study will assess the feasibility of the workflow. A subset of participants will be re-contacted at 3 months to evaluate referral completion and retention rates. The ultimate goal is to establish a non-stigmatizing, objective triage protocol to improve mental health resource utilization in digestive clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 60 years, regardless of sex.
2. Diagnosed with chronic atrophic gastritis (CAG) confirmed by upper gastrointestinal endoscopy and histopathology within the past 6 months.
3. Ability to comprehend and voluntarily complete psychological assessments and multimodal vascular examinations.
4. Willingness to provide written informed consent.

Exclusion Criteria:

1. History of major psychiatric disorders (e.g., schizophrenia, bipolar disorder) or currently experiencing an acute psychotic episode.
2. Major cardiovascular or cerebrovascular events (e.g., acute myocardial infarction, stroke) within the past 3 months.
3. Severe peripheral artery disease or major anatomical abnormalities in the lower extremities (e.g., Fontaine stage III-IV, diabetic foot with ulcers) that would preclude reliable dorsalis pedis artery ultrasound assessment.
4. Severe hepatic or renal dysfunction, or malignancy with a limited life expectancy.
5. Current use of systemic corticosteroids or potent immunosuppressants.
6. Pregnancy or lactation.
7. Any other condition deemed by the investigators to interfere with study participation or cooperation.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of adult patients (aged 20-60 years) with histologically confirmed chronic atrophic gastritis (CAG). Participants are recruited from the gastroenterology outpatient clinics of four participating centers in Northern and Eastern China (including China Academy of Chinese Medical Sciences, Beijing Anzhen Hospital, Hengshui Hospital of TCM, and Liyang Hospital of TCM). All participants must have undergone upper gastrointestinal endoscopy within the past 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptom Screening-Positive Status (PHQ-9 ≥10) | Baseline (Day 0)
  The primary outcome is the binary classification of depressive symptom burden. Participants are categorized as "screen-positive" if their 9-item Patient Health Questionnaire (PHQ-9) total score is ≥10, indicating moderate-to-severe depressive symptoms warranting referral. The PHQ-9 scores range from 0 to 27, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Screening Completion Rate | Up to 3 months
  The proportion of eligible patients consenting to assessment.
Referral Uptake Rate | Up to 3 months
  The proportion of screen-positive patients completing mental health consultation.
Dorsalis Pedis Artery Resistive Index (RI) | Baseline (Day 0)
  A calculated flow parameter reflecting vascular resistance measured via Doppler ultrasound.
Dorsalis Pedis Artery Pulsatility Index (PI) | Baseline (Day 0)
  A calculated flow parameter reflecting vascular pulsatility measured via Doppler ultrasound.
Dorsalis Pedis Artery Flow Waveform Classification | Baseline (Day 0)
  Flow waveforms classified into three categories: triphasic, biphasic, or monophasic via Doppler ultrasound assessment.
Brachial-Ankle Pulse Wave Velocity (baPWV) | Baseline (Day 0)
  Measured to assess arterial stiffness.
Generalized Anxiety Disorder-7 (GAD-7) Score | Baseline (Day 0)
  Anxiety symptom severity assessed using the GAD-7 scale. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Time Burden | Up to 3 months
  The median time added to routine workflow (measured in minutes)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Hengshui Hospital of Traditional Chinese Medicine, Hengshui, Hebei
  - Liyang Hospital of Chinese Medicine, Changzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification, may be shared with researchers who provide a methodologically sound proposal and obtain necessary ethical approvals. Data sharing is subject to the rules and regulations of the participating institutions and the Data Security Law of China.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to the corresponding author (wangchao19891216@163.com). To gain access, data requestors will need to sign a data access agreement and provide ethical approval from their institution.